CLINICAL TRIAL: NCT00335647
Title: A Phase I/IIa, Open-Label, Dose-Escalation Study to Determine the Safety, Tolerance, and Preliminary Activity of Intravenous High-Dose Fluphenazine HCI in Patients With Advanced Multiple Myeloma
Brief Title: Fluphenazine in Treating Patients With Refractory Advanced Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immune Control (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000486281; IMMUNECON-FM-CL1; UPCC-IRB-5; UPCC-09405; UPCC-803972
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage III multiple myeloma; refractory multiple myeloma; stage II multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Fluphenazine

INTERVENTIONS:
Drug: fluphenazine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluphenazine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of fluphenazine and to see how well it works in treating patients with refractory advanced multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of high-dose fluphenazine hydrochloride in patients with refractory advanced multiple myeloma.
* Determine the pharmacological properties of this drug.
* Determine the effectiveness of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive high-dose fluphenazine hydrochloride IV 3 times on day 1. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive escalating doses of fluphenazine hydrochloride until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed multiple myeloma

  * Advanced disease
  * Must be refractory to ≥ 2 different methods of standard treatment
* Measurable disease, defined as serum paraprotein ≥ 1g/L or urine light chain ≥ 200 mg/24 hours
* No brain involvement or leptomeningeal disease
* No spinal cord compression unless the following criteria are met:

  * Patient has undergone prior surgery or radiotherapy
  * Neurological findings are ≤ grade 1
  * Patient is off steroids for spinal cord edema or is on a stable regimen of ≤ 10 mg/day of prednisone or equivalent

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 (ECOG PS 3 allowed if related to skeletal lesions)
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,000/mm^3*
* Platelet count ≥ 50,000/mm^3*
* Hemoglobin ≥ 8.0 g/dL* (no transfusion within the past 7 days)
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* Creatinine clearance ≥ 30 mL/min
* LVEF ≥ 40%
* QTc < 450 msec
* No evidence of dysrhythmias on EKG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No congestive heart failure
* No angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 180 mm Hg and/or diastolic BP > 105 mm Hg
* No myocardial infarction within the past year
* No active infection
* No HIV, hepatitis B, or hepatitis C infection
* No history of psychosis
* No history of subcortical brain damage
* No hypersensitivity to fluphenazine hydrochloride or other phenothiazines
* No history of seizures or extrapyramidal symptoms
* No other serious illness or medical condition
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix NOTE: *Patients with values outside of this range due to infiltration by myeloma may be allowed at the discretion of the investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 21 days since prior chemotherapy, immunotherapy, or radiotherapy
* At least 21 days since prior and no concurrent systemic steroids

  * Patients who have been taking chronically administered steroids for ≥ 1 month at a dose ≤ 10 mg/day of prednisone or equivalent are eligible
* At least 28 days since prior investigational agents
* At least 6 weeks since prior selective serotonin reuptake inhibitors (SSRIs) (a wash-out period equivalent to 5 times the terminal elimination half-life is required for tricyclic antidepressants or norepinephrine reuptake inhibitors)
* No concurrent SSRIs, tricyclic antidepressants, or norepinephrine reuptake inhibitors
* No concurrent dialysis therapy
* No concurrent hematopoietic growth factors except epoetin alfa

  * Treatment with hematopoietic growth factors may be started during study if patient develops or has progressive cytopenia
* No concurrent anticholinergics or other antipsychotics
* No concurrent antiseizure drugs except Neurontin for treatment of neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania